CLINICAL TRIAL: NCT07190482
Title: Treatment of Tinnitus With Olanzapine: A Randomized Crossover Versus Placebo Study
Brief Title: Treatment of Tinnitus With Olanzapine
Acronym: OLANZAP_TIN
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Sao Paulo (Other)
Responsible Party: Principal Investigator, Jeanne Oiticica, MD PhD, University of Sao Paulo
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 6.414.085
Record Dates: First submitted 2025-09-12; First posted 2025-09-24 (Actual); Last update posted 2025-09-24 (Actual); Status verified 2025-09

CONDITIONS: Tinnitus; Tinnitus, Subjective
Keywords: TINNITUS; OLANZAPINE
MeSH Terms: conditions — Tinnitus | interventions — Olanzapine; Tablets

STUDY DESIGN:
Intervention Model Description: To evaluate the efficacy of olanzapine in reducing tinnitus symptoms in a randomized placebo-controlled crossover trial
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- OLANZAPINE ARM (Active Comparator): olanzapine 5 mg/day administered for 8 weeks
  Interventions: Drug: Olanzapine 5 Mg ORAL TABLET
- PLACEBO ARM (Placebo Comparator): placebo administered for 8 weeks
  Interventions: Drug: Placebo Drug

INTERVENTIONS:
Drug: Olanzapine 5 Mg ORAL TABLET — OLANZAPINE ARM
  Other Names: Zyprexa; OLZ
  Arms: OLANZAPINE ARM
Drug: Placebo Drug — placebo administered for 8 weeks
  Other Names: Sham treatment
  Arms: PLACEBO ARM

SUMMARY:
This research aims to evaluate the effects of the drug olanzapine on the discomfort caused by tinnitus according to each patient's personality traits. Olanzapine is a drug used as an antipsychotic whose mechanism of action makes it potentially useful for the treatment of tinnitus.

DETAILED DESCRIPTION:
Patients will be evaluated through a standard history and otorhinolaryngological examination. Questionnaires will be used to assess tinnitus (Tinnitus Handicap Inventory) and personality (Neo Pi-R), and audiological examinations will be performed (pure-tone and vocal audiometry and immittance testing). All procedures aim to understand the impact of the disease on the patient's life, and audiological examinations aim to analyze the patient's hearing. To perform the procedures and examinations and monitor the treatment schedule, the patient will be required to attend the outpatient clinic monthly. The procedures and examinations do not pose any risk or physical discomfort to the interviewee.

ELIGIBILITY:
Inclusion Criteria:

* Subjective, non-pulsatile tinnitus of at least 6 months' duration
* Stable tinnitus symptoms over the past 3 months
* Willingness to participate and provide informed consent
* Age between 18 and 70 years

Exclusion Criteria:

* Active psychiatric disorders requiring pharmacological treatment
* History of psychotic illness or bipolar disorder
* Current use of antipsychotics, antidepressants, or anticonvulsants
* Severe hearing loss (threshold ≥ 80 dB in both ears)
* Substance use disorders
* Pregnancy or breastfeeding
* Known hypersensitivity to olanzapine
* Significant medical conditions (e.g., uncontrolled diabetes, hepatic impairment)

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2023-10-01 (Actual); Primary Completion 2024-12-20 (Actual); Study Completion 2025-01-20 (Actual)

PRIMARY OUTCOMES:
Evaluate the efficacy of olanzapine in reducing tinnitus symptoms in a randomized placebo-controlled crossover trial | From enrollment to the end of treatment at 12 weeks
  • Tinnitus Handicap Inventory (THI): A 25-item questionnaire measuring tinnitus-related distress. Scores range from 0 to 100, with higher scores indicating greater handicap.

SECONDARY OUTCOMES:
Assess the clinical efficacy of olanzapine (5 mg/day) in reducing tinnitus symptoms, using a randomized, double-blind, placebo-controlled crossover design | From enrollment to the end of treatment at 12 weeks
  • Visual Analog Scales (VAS): Patients rated tinnitus loudness and distress on 10-point scales (0 = none; 10 = extreme).

CONTACTS AND LOCATIONS:
Overall Officials: Research Ethics Committee (CEP) Research Ethics Committee (CEP), Principal Investigator — Research Ethics Committee (CEP); JEANNE OITICICA, MD PhD, Study Chair — Research Ethics Committee (CEP)
Locations (1):
- Research Ethics Committee (CEP), São Paulo, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No